CLINICAL TRIAL: NCT06104098
Title: A User Study With Vernivia® for Bacterial Vaginosis (USV01) Evaluation of User-friendliness, Measure Time From the Start of Treatment to Symptom Relief and the Clarity of Instructional Material
Brief Title: A User Study With Vernivia® for Bacterial Vaginosis.
Acronym: USV01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepTonic Medical AB (Industry)
Collaborators: Key2Compliance (Industry); Replior AB (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USV01
Record Dates: First submitted 2021-09-02; First posted 2023-10-27 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Bacterial Vaginoses
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One dose daily for 7 consequtive days (dose acc to IFU) (Other): Open user study with Vernivia once daily for 7 consequtive days. Dosage according to IFU/Instructions For Use.
  Interventions: Device: D005 vaginal mousse

INTERVENTIONS:
Device: D005 vaginal mousse — D005 Vaginal Mousse is class IIa medical device for treatment of Bacterial Vaginosis.
  Other Names: Vernivia

SUMMARY:
This is an open user study to evaluate D005 vagnial mousse with regards to user-friendliness, and measure time from start of treatment to symptom relief and measure the clarity of instructional material.

The study will be conducted at seven sites in Sweden, the study population will consist of up to 100 female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 - 49 years Informed consent to take part in the study Bacterial vaginosis (based on self-assessment or diagnosed by a doctor or midwife) Access to a smartphone

Exclusion Criteria:

* Symptoms of vaginal candida infection and/or Pregnancy

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
Evaluate symptom relief during treatment with Vernivia®. | 1-7 days
  Evaluation of number of days from start of treatment until symptom relief

SECONDARY OUTCOMES:
Self-reported grading of malodorous discharge (0-3) | 1-7 days
  Evaluate how the user experiences the product with regards to malodorous
  (1 = Not likely, 10 = Very likely)
Net Promotor Score regarding user-friendliness | 1-7 days
  Evaluate how the user experiences the user-friendliness
  (1 = Not likely, 10 = Very likely)
Clarity of the IFU (Instructions For Use) | 1-7 days
  Evaluate how the user experiences the IFU (Instructions For Use)
  (1= Not at all informative, 5= Very informative)
Clarity of instructional video | 1-7 days
  Evaluate how the user experiences the instructional video
  (1= Not at all informative, 5= Very informative)

CONTACTS AND LOCATIONS:
Locations (7):
- Sweden (7):
  - Mama Mia Väla, Väla, Helsingborg
  - Mednika AB, Linköping
  - Hälsomedicinskt Center, Lomma
  - Mama Mia Barnmorskemottagning, Malmo
  - Kvinnohälsan Stadsfjärden, Nyköping
  - 2Heal Medical, Stockholm
  - Ondrasek Läkarmottagning, Sundsvall

IPD SHARING:
Plan to Share IPD: No